CLINICAL TRIAL: NCT05350800
Title: A Phase 1, Two-part Study to Evaluate the Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of BMS-986369 and to Explore the Effect of Food the Bioavailability of BMS-986369 in Healthy Participants
Brief Title: A Study to Evaluate the Drug Exposure of Single Ascending Doses of BMS-986369 and the Effect of Food on the BMS-986369 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA073-001
Record Dates: First submitted 2022-04-25; First posted 2022-04-28 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer
Keywords: BMS-986369; Healthy Volunteer; CC-99282

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986369, Part 1 dose escalation (Experimental)
  Interventions: Drug: BMS-986369
- BMS-986369 under fasted conditions, Part 2 Food effect (Experimental)
  Interventions: Drug: BMS-986369
- BMS-986369 under fed conditions, Part 2 Food effect (Experimental)
  Interventions: Drug: BMS-986369

INTERVENTIONS:
Drug: BMS-986369 — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels of BMS-986369 following administration of single ascending oral doses (SAD) in healthy adult participants. The study will also explore the effect of high-fat meal on the single-dose drug level of BMS-986369 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.0 to 33.0 kg/m2, inclusive. BMI = weight (kg)/(height [m])2 for participants
* Must have a normal or clinically-acceptable 12-lead ECG at screening
* Absolute neutrophil counts must be greater than 2,500/μL at screening and Day -1

Exclusion Criteria:

* Any significant acute or chronic medical illness that presents a potential risk to the participant in the opinion of the investigator and/or may compromise the objectives of the study
* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular (CV), peripheral vascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary (GU) abnormalities/diseases
* History of major surgery within 8 weeks before the first dose administration

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1
Time of maximum observed plasma concentration (Tmax) | Day 1
Area under the plasma concentration-time curve, from time zero extrapolated to infinite time (AUC(INF)) | Up to 336 hours after dose administration

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From the date of having consented until 30 days after completion of study treatment
Number of participants with vital sign abnormalities | Up to Day 15
Number of participants with clinical laboratory abnormalities | Up to Day 15
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 15
Effect of BMS-986369 on ECG parameters - Part 1 | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT05350800.html